CLINICAL TRIAL: NCT06126276
Title: A Randomized Trial of Neratinib, A Pan-ERBB Inhibitor, Alone or in Combination With Palbociclib, a CDK4/6 Inhibitor, in Patients With HER2+ Gynecologic Cancers and Other Solid Tumors: A ComboMATCH Treatment Trial
Brief Title: Testing the Use of Neratinib or the Combination of Neratinib and Palbociclib Targeted Treatment for HER2+ Solid Tumors (A ComboMATCH Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-09270; NCI-2023-09270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-N5 (Other: NRG Oncology); EAY191-N5 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Malignant Female Reproductive System Neoplasm; Malignant Solid Neoplasm; Recurrent Malignant Female Reproductive System Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; neratinib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (neratinib maleate) (Active Comparator): Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may crossover to Arm II. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Neratinib Maleate
- Arm II (neratinib maleate, palbociclib) (Experimental): Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 and palbociclib PO QD on days 1-21 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Neratinib Maleate; Drug: Palbociclib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Neratinib Maleate — Given PO
  Other Names: 2-Butenamide, N-(4-((3-chloro-4-(2-pyridinylmethoxy)phenyl)amino)-3-cyano-7-ethoxy-6-quinolinyl)-4-(dimethylamino)-, (2E)-, (2Z)-2-butenedioate (1:1); HKI-272 Maleate; NERATINIB MALEATE ANHYDROUS; Nerlynx
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991
  Arms: Arm II (neratinib maleate, palbociclib)

SUMMARY:
This phase II ComboMATCH treatment trial compares the effect of neratinib to the combination of neratinib and palbociclib in treating patients with HER2 positive solid tumors. Neratinib and palbociclib are in a class of medications called kinase inhibitors. They work by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of tumor cells. Giving neratinib and palbociclib in combination may shrink or stabilize cancers that over-express a specific biomarker called HER2.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the efficacy of neratinib plus palbociclib (PD-0332991) compared to neratinib maleate (neratinib) alone in patients with HER2+ gynecologic cancers and HER2+ solid tumors by evaluating progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. To investigate outcome in terms of objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To investigate clinical benefit rate (ORR + stable disease at 16 weeks). III. To evaluate overall (OS) survival. IV. To evaluate the ORR of patients who crossed over from neratinib monotherapy to neratinib-palbociclib combination.

V. To investigate adverse events especially grade 3 and 4 toxicities by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

VI. Collect tissue and provide it to the ComboMATCH Registration Protocol to assess concordance between the diagnostic tumor mutation profile generated by the Designated Laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor-derived deoxyribonucleic acid (ctDNA) mutation profile from plasma, as described in ComboMATCH Registration Protocol.

EXPLORATORY TRANSLATIONAL OBJECTIVES:

I. To investigate the role of ctDNA-HER2 status at baseline and during follow up to assess if it predicts response to therapy and disease progression and if it does correlate with tumor tissue based HER2 status.

II. To investigate if activation of the pathways of interest (PI3K/mTOR and RB1, CCND1-CDK4/6 CDK and RAS/RAF/MAPK) in tumor tissue as well as blood/ctDNA correlate with response or resistance to therapy.

III. To correlate extent of HER2 amplification with response to treatment and with HER2 expression by immunohistochemistry or fluorescence in situ hybridization (FISH).

IV. To correlate the extent of HER2 amplification with HER2 expression by RNA and protein immunohistochemistry (IHC) analyses and FISH.

V. To correlate expression of Rb1, CCND1, CCNE1, CDK4/6 protein expression with response to treatment.

VI. Assess alteration in RB1-CDK pathway in neratinib resistant patients at time of progression on monotherapy compared to combination neratinib-palbociclib.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive neratinib maleate orally (PO) once daily (QD) on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may crossover to Arm II. Patients undergo echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) during screening and on study, and computed tomography (CT) or magnetic resonance imaging (MRI) and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.

ARM II: Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 and palbociclib PO QD on days 1-21 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-N5 based on the presence of an actionable mutation as defined in EAY191
* Patients must have a HER2 amplified solid tumor except breast cancer.

  * If IHC is 0 or 1+, patient (pt) is NOT ELIGIBLE regardless of FISH or next generation sequencing (NGS) status
  * If IHC is 3+, pt IS ELIGIBLE regardless of FISH or NGS status
  * If IHC is 2+, FISH OR NGS must be positive for the patient to be ELIGIBLE. Otherwise, pt is NOT ELIGIBLE
  * If IHC is unknown and…

    * FISH is positive, independent of NGS results, the patient IS ELIGIBLE
    * FISH is negative and NGS positive with ≥7 copies, the patient IS ELIGIBLE
* Patients must have recurrent or persistent disease
* No known evidence of RB1 loss or deletion including copy number loss or deleterious mutation
* Patients must have disease that can be safely biopsied and agree to a pre-treatment biopsy or, if disease cannot be safely biopsied, have archival tissue available from within 12 months prior to the date of registration on the ComboMATCH Registration Trial (EAY191)
* Patients must have measurable disease based on RECIST 1.1. A second measurable lesion outside of the biopsiable lesion is required
* Patients with treated brain metastases are eligible if follow up brain imaging after central nervous system (CNS) directed therapy shows no evidence of progression for 3 months or more and patient is not on steroids and is asymptomatic
* No known leptomeningeal disease
* Patients may have received up to 5 prior lines of systemic therapy
* Prior therapy with trastuzumab or pertuzumab, either alone or in combination, antibody drug conjugates (ADC) such as DS8201a or T-DM1 is allowed
* Prior therapy with tyrosine kinase inhibitors (TKI) such as neratinib or tucatinib is not allowed
* No prior therapy with CDK4/6 inhibition
* No cancer directed therapy within 3 weeks prior to registration. For oral therapy, the washout can be reduced to greater than or equal to 5 half lives of the drug. No HER2 targeting ADCs within 30 days prior to registration
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Not pregnant and not nursing
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 9 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin (Hgb) ≥ 9 g/dl is acceptable)
* Creatinine clearance (CrCL) of ≥ 30 mL/min by the Cockcroft-Gault formula
* Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level ≤ 3 x institutional ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional upper limit of normal (ULN)
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* No active infection requiring parenteral antibiotics
* No current evidence of intra-abdominal abscess, abdominal/pelvic fistula (not diverted), gastrointestinal perforation, gastrointestinal (GI) obstruction, and/or need for drainage nasogastric or gastrostomy tube
* No current evidence of malabsorption or chronic diarrhea or any other significant gastro-intestinal disease (e.g gastrectomy, ileal bypass, Crohn's disease, gastroparesis), associated with moderate to severe diarrhea (grade 2 or more) or inability to tolerate oral therapy
* No lung disease causing dyspnea at rest
* No interstitial lung disease with ongoing signs and symptoms at the time of registration
* No history of allergic reaction to the study agents, compound of similar chemical or biologic composition of the study agents or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 2 years
  The stratified log-rank statistic will be used to draw inferences about the relative activity of the two regimens. Characterized by medians and Kaplan-Meier (KM) curves.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  The impact of treatment on the hazard of death can be investigated with time dependent covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Haider S Mahdi, Principal Investigator — NRG Oncology
Locations (180):
- United States (180):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - SIH Cancer Institute, Carterville, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Mercyhealth Cancer Institute - Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Woodland Cancer Care Center, Michigan City, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Regional Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.html